CLINICAL TRIAL: NCT01978704
Title: Use of the Glycemic Load for the Adjustment of the Dose of Preprandial Insulin in Patients With Type 1 Diabetes Mellitus in Insulin Pump Therapy
Brief Title: Glycaemic Load and Pre-meal Insulin Doses in Type 1 Diabetes Patients
Acronym: GLUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Prof, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 37/13
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycaemic load (Experimental)
  Interventions: Other: Adjustment of pre-prandial insulin doses on the bases of glycaemic load of the meal
- Carbohydrates content (Active Comparator)
  Interventions: Other: Adjustment of pre-prandial insulin doses on the bases of carbohydrates content of the meal

INTERVENTIONS:
Other: Adjustment of pre-prandial insulin doses on the bases of glycaemic load of the meal
  Arms: Glycaemic load
Other: Adjustment of pre-prandial insulin doses on the bases of carbohydrates content of the meal
  Arms: Carbohydrates content

SUMMARY:
The aim of this study is to compare the feasibility and the efficacy on short-term glucose control of pre-meal insulin doses adjustment made on the bases of the glycemic load or of the carbohydrates content of the meal in patients with type 1 diabetes mellitus treated with insulin pump

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes treated by insulin pump

Exclusion Criteria:

* Preganncy
* HbA1c > 9%

  * Any serious acute or chronic illness a part diabetes

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
daily plasma glucose excursion | 1 week
mean plasma glucose concentrations | 1 week

SECONDARY OUTCOMES:
postprandial plasma glucose concentrations | 1 week